CLINICAL TRIAL: NCT01179334
Title: An Interaction Study to Evaluate Changes in Blood Pressure Following 1, 1.5, 2, and 2.5 mg Riociguat Tid (Dose Titration) Compared to Placebo Treatment on the Background of Stable Sildenafil Pretreatment in Subjects With Symptomatic Pulmonary Arterial Hypertension
Brief Title: Evaluation of the Pharmacodynamic Effect of the Combination of Sildenafil and Riociguat on Blood Pressure and Other Safety Parameters.
Acronym: PATENT PLUS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 15096; 2010-018863-40 (EudraCT Number)
Record Dates: First submitted 2010-08-10; First posted 2010-08-11 (Estimated); Results first posted 2013-12-25 (Estimated); Last update posted 2016-08-29 (Estimated); Status verified 2016-07

CONDITIONS: Pulmonary Hypertension
Keywords: Pulmonary Hypertension; Riociguat; Blood Pressure
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — riociguat; Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Riociguat (Adempas, BAY63-2521) up to 2.5 mg_IDT (Experimental): Participants received Riociguat orally as a film-coated tablet up to 2.5mg three times daily (tid) (titration between 1.0 mg and 2.5 mg tid based on an individual dose titration (IDT) scheme) for 12 weeks. Participants continued to take daily stable sildenafil background treatment according to their prescriptions.
  Interventions: Drug: Riociguat (Adempas, BAY63-2521); Drug: Sildenafil
- Placebo (Placebo Comparator): Participants received Placebo orally as a film-coated tablet three times daily (tid) for 12 weeks. Participants continued to take daily stable sildenafil background treatment according to their prescriptions.
  Interventions: Drug: Placebo; Drug: Sildenafil

INTERVENTIONS:
Drug: Riociguat (Adempas, BAY63-2521) — BAY63-2521: 1 mg tid - 2,5 mg tid oral for 12 weeks.
  Arms: Riociguat (Adempas, BAY63-2521) up to 2.5 mg_IDT
Drug: Placebo — Placebo for 12 weeks
  Arms: Placebo
Drug: Sildenafil — Participants continued to take daily stable sildenafil background treatment according to their prescriptions.

SUMMARY:
Pulmonary Arterial Hypertension (PAH) is a severe progressive disease with a high mortality. Although several drugs are available for the treatment of PAH none offer a cure, therefore there is still a high medical need for new treatments.

Soluble guanylate cyclase (sGC) is one of the chemicals involved in the pathways controlling vascular tone, which is impaired in patients with PAH. This causes constriction and thickening of the blood vessels wall in the lungs and increase of blood pressure in the lungs. This can lead to the very debilitating symptoms of PAH such as tiredness, shortness of breath on exertion, collapse and often the inability of the patient to perform their daily life activities.

Inhalation of Nitric Oxide, which activates sGC is used to treat PAH, but its effect wears off as soon as inhalation stops. Direct stimulation of sGC using this new compound Riociguat may be a new approach for the treatment of PAH.

The phosphodiesterase 5 (PDE5)-inhibitor Sildenafil is one of licensed treatments for PAH. The Patent Plus is a double-blind, placebo-controlled safety study, designed to investigate the effect of Riociguat on blood pressure in patients with PAH when given in combination with Sildenafil.

DETAILED DESCRIPTION:
Main objective: Evaluation of the pharmacodynamic effect of the combination of Sildenafil and Riociguat on blood pressure and other safety parameters in patients with symptomatic PAH Secondary objectives:To investigate the safety of the riociguat/sildenafil combination and changes in 6-minute walk test, World Health Organization (WHO) functional class, N terminal pro-brain natriuretic peptide, and variables obtained during right-heart catheterization after 12 weeks of treatment; pharmacokinetics of riociguat and sildenafil.

The study consists of one part. In study Part 1 only subjects (18) on stable sildenafil treatment of 20 mg tid have been enrolled. Study Part 2 will not start.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 75 years of age at Visit 1
* Male and female subjects with symptomatic PAH (Group I Dana Point Updated Clinical Classification 2008), a 6-min walking distance (6MWD) of more than 150 m, a pulmonary vascular resistance (PVR) >300 dyn*s*cm-5, and a mean pulmonary artery pressure (PAPmean) ≥ 25 mmHg
* For Study Part 1: subjects on stable pretreatment with sildenafil at a dose of 20 mg tid
* Unspecific treatments which may also be used for the treatment of PAH such as oral anticoagulants, diuretics, digitalis, calcium channel blockers or oxygen supplementation are permitted. However, treatment with anticoagulants (if indicated) must have been started at least 30 days before Visit 1 and treatment with diuretics needs to be stable for at least 30 days before Visit 1
* Subjects with supplemental long-term oxygen therapy may be included, if the amount of supplemental oxygen and the delivery method was stable on average for at least 90 days before Visit 1
* SBP >/=95 mmHg and heart rate (HR) </=105 beats per minute (BPM) in the first 2 h after intake of sildenafil (measured at Visits 0 and 1)
* Women without child-bearing potential
* Subjects who are able to understand and follow instructions and who are able to participate in the study for the entire period
* Subjects must have given their written informed consent to participate in the study after having received adequate previous information and prior to any study-specific procedures

Exclusion Criteria:

* Subject's participating in another clinical trial or who have done so within 30 days before Visit 1
* Previous assignment to treatment during this study
* Pregnant women
* Subjects with a medical disorder, condition, or history of such that would impair the subject's ability to participate or complete this study in the opinion of the investigator
* Subjects with substance abuse (eg alcohol or drug abuse) within the previous 180 days before Visit 1
* Subjects with underlying medical disorders with an anticipated life expectancy below 2 years (eg active cancer disease with localized and/or metastasized tumor mass)
* Subjects with a history of severe allergies or multiple drug allergies
* Subjects with hypersensitivity to the investigational drug or any of the excipients
* Subjects unable to perform a valid 6MWD test, eg subjects with a severe peripheral artery occlusive disease
* Subjects with a relative difference (ie absolute difference/mean) of more than 15% between the eligibility- and the baseline 6MWD test
* All types of pulmonary hypertension except subtypes of Updated Clinical Classification of pulmonary hypertension (PH) (Dana Point 2008) Group I specified in the inclusion criteria
* Moderate to severe obstructive lung disease (forced expiratory volume <60% predicted). The predicted forced expiratory volume in 1 second (FEV1) is a calculated value
* Severe restrictive lung disease (total lung capacity <70% predicted). The predicted total lung capacity (TLC) is a calculated value
* Severe congenital abnormalities of the lungs, thorax, and diaphragm
* Oxygen saturation (SaO2) <88% despite supplemental oxygen therapy
* Arterial partial oxygen pressure (PaO2) <55 mmHg despite supplemental oxygen therapy
* Arterial partial pressure of carbon dioxide (PaCO2) >45 mmHg
* Uncontrolled arterial hypertension (SBP >180 mmHg and /or diastolic blood pressure >110 mmHg
* Atrial fibrillation within the last 90 days before Visit 1
* Pulmonary venous hypertension with pulmonary capillary wedge pressure 15 mmHg
* Hypertrophic obstructive cardiomyopathy
* Severe proven or suspected coronary artery disease
* Clinical evidence of symptomatic atherosclerotic disease
* Congenital or acquired valvular or myocardial disease if clinically significant apart from tricuspid valvular insufficiency due to pulmonary hypertension
* Clinical relevant hepatic dysfunction indicated by:

  * Bilirubin >2 times upper limit normal (ULN)
  * and/or ALT (alanine aminotransferase) or AST (aspartate aminotransferase) >3 times ULN
  * and/or signs of severe hepatic insufficiency (eg impaired albumin synthesis with an albumin <32 g/L, hepatic encephalopathy > grade 1
* Renal insufficiency (glomerular filtration rate <30 mL/min, eg calculated based on the Cockcroft-Gault or Modification of Diet in Renal Disease (MDRD) formulas

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2010-08; Primary Completion 2012-06 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (25):
- United States (3):
  - Aurora, Colorado
  - Columbus, Ohio
  - Providence, Rhode Island
- Austria (2):
  - Innsbruck
  - Villach
- Vseobecna fakultni nemocnice, Prague, Czechia
- Germany (10):
  - Heidelberg, Baden-Wurttemberg
  - Regensburg, Bavaria
  - Würzburg, Bavaria
  - Hamburg, Hamburg
  - Giessen, Hesse
  - Hanover, Lower Saxony
  - Cologne, North Rhine-Westphalia
  - Mönchengladbach, North Rhine-Westphalia
  - Dresden, Saxony
  - Berlin, State of Berlin
- Italy (2):
  - Bologna, Emilia-Romagna
  - Pavia, Lombardy
- New Zealand (2):
  - Auckland
  - Christchurch
- Poland (2):
  - Otwock
  - Warsaw
- Barcelona, Barcelona, Spain
- United Kingdom (2):
  - Papworth Hospital, Cambridge, Cambridgeshire
  - Clydebank, West Dunbartonshire

REFERENCES:
- [Result] Galie N, Muller K, Scalise AV, Grunig E. PATENT PLUS: a blinded, randomised and extension study of riociguat plus sildenafil in pulmonary arterial hypertension. Eur Respir J. 2015 May;45(5):1314-22. doi: 10.1183/09031936.00105914. Epub 2015 Feb 5. PMID 25657022

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Only participants with symptomatic Pulmonary arterial hypertension (PAH) could participate in this study. Subjects must be on pre-treatment with sildenafil at a dose of 20 mg three times daily (tid) (20 or 25 mg tid in New Zealand) for at least 90 days.
Pre-assignment Details: 24 subjects were enrolled in 11 study centers in 5 European countries. Six of the 24 subjects were screened but not randomized (screen failure [6]). 18 of the 24 participants were randomized. All of the 18 randomized participants received study medication.
Period: Treatment Period
Arm/Group | Riociguat (Adempas, BAY63-2521) up to 2.5 mg_IDT | Placebo
Started | 12 | 6
Participants Received Treatment | 12 | 6
Completed | 11 | 6
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Long-term Extension (LTE) Period
Arm/Group | Riociguat (Adempas, BAY63-2521) up to 2.5 mg_IDT | Placebo
Started | 11 | 6
Completed | 0 (LTE phase was terminated by sponsor) | 0 (LTE phase was terminated by sponsor)
Not Completed | 11 | 6
Not completed — Study terminated by sponsor | 6 | 2
Not completed — Death | 3 | 0
Not completed — Adverse Event | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Riociguat (Adempas, BAY63-2521) up to 2.5 mg_IDT | Placebo | Total
Number analyzed (Participants) | 12 | 6 | 18
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.3 (10.7) | 61.3 (10.0) | 59.3 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 12
  Male | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Maximum Change From Baseline in Supine Systolic Blood Pressure (SBP) Within 4 Hours Post-dose at Visit 6 (Week 12)
Description: Systolic blood pressure (SBP) was measured as standard vital sign parameter. Range allowed in this study: <= 180 mmHg. In addition, SBP must be >=95 mmHg in the first 2 hours after intake of background treatment with sildenafil. The maximum change from baseline at each visit was defined as the within-subject maximum decrease from baseline (or zero if baseline was lower than all subsequent SBP measurements in that profile) within 4 hours post-dose. Baseline was the last SBP recorded at and within 30 minutes before intake of study drug.
Time Frame: Pre-dose (baseline) and within 4 hours post-dose at visit 6 (week 12)
Population: pharmacodynamic(s) (PD) analysis set
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Riociguat (Adempas, BAY63-2521) up to 2.5 mg_IDT | Placebo
Number analyzed (Participants) | 10 | 5
mmHg | -20.70 (17.97) | -20.20 (12.91)

2. Secondary Outcome: Maximum Change From Baseline in Standing Systolic Blood Pressure (SBP) Within 4 Hours Post-dose at Visit 6 (Week 12)
Description: as for outcome 1
Time Frame: Pre-dose (baseline) and within 4 hours post-dose at visit 6 (week 12)
Population: PD analysis set
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Riociguat (Adempas, BAY63-2521) up to 2.5 mg_IDT | Placebo
Number analyzed (Participants) | 10 | 5
mmHg | -18.00 (16.50) | -16.80 (10.62)

3. Secondary Outcome: Maximum Change From Baseline in Supine Diastolic Blood Pressure (DBP) Within 4 Hours Post-dose at Visit 6 (Week 12)
Description: Diastolic blood pressure (DBP) was measured as standard vital sign parameter. Range allowed in this study: <= 110 mmHg. The maximum change from baseline at each visit was defined as the within-subject maximum decrease from baseline (or zero if baseline was lower than all subsequent DBP measurements in that profile) within 4 hours post-dose. Baseline was the last DBP recorded at and within 30 minutes before intake of study drug.
Time Frame: Pre-dose (baseline) and within 4 hours post-dose at visit 6 (week 12)
Population: PD analysis set
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Riociguat (Adempas, BAY63-2521) up to 2.5 mg_IDT | Placebo
Number analyzed (Participants) | 10 | 5
mmHg | -13.70 (11.72) | -13.80 (12.85)

4. Secondary Outcome: Maximum Change From Baseline in Standing Diastolic Blood Pressure (DBP) Within 4 Hours Post-dose at Visit 6 (Week 12)
Description: as for outcome 3
Time Frame: Pre-dose (baseline) and within 4 hours post-dose at visit 6 (week 12)
Population: PD analysis set
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Riociguat (Adempas, BAY63-2521) up to 2.5 mg_IDT | Placebo
Number analyzed (Participants) | 10 | 5
mmHg | -14.40 (10.59) | -14.20 (10.03)

5. Secondary Outcome: Maximum Change From Baseline in Supine Heart Rate (HR) Within 4 Hours Post-dose at Visit 6 (Week 12)
Description: Heart rate (HR) was measured as standard vital sign parameter. Range allowed in this study: <= 105 beats per minute (bpm) in the first 2 hours after intake of background treatment with sildenafil. The maximum change from baseline at each visit was defined as the within-subject maximum increase from baseline (or zero if baseline was higher than all subsequent HR measurements in that profile) within 4 hours post-dose. Baseline was the last HR recorded at and within 30 minutes before intake of study drug.
Time Frame: Pre-dose (baseline) and within 4 hours post-dose at visit 6 (week 12)
Population: PD analysis set
Measure: Mean (Standard Deviation); unit: Beats/min
Arm/Group | Riociguat (Adempas, BAY63-2521) up to 2.5 mg_IDT | Placebo
Number analyzed (Participants) | 10 | 5
Beats/min | 5.90 (7.14) | 9.60 (5.50)

6. Secondary Outcome: Maximum Change From Baseline in Standing Heart Rate (HR) Within 4 Hours Post-dose at Visit 6 (Week 12)
Description: as for outcome 5
Time Frame: Pre-dose (baseline) and within 4 hours post-dose at visit 6 (week 12)
Population: PD analysis set
Measure: Mean (Standard Deviation); unit: Beats/min
Arm/Group | Riociguat (Adempas, BAY63-2521) up to 2.5 mg_IDT | Placebo
Number analyzed (Participants) | 10 | 5
Beats/min | 6.50 (7.17) | 10.40 (6.54)

7. Secondary Outcome: Area Under Effect Curve (AUEC) of Supine SBP Within 4 Hours Post-dose at Visit 6 (Week 12)
Description: The area under the effect curve (AUEC) at each visit of supine SBP describes an average within-subject change in SBP from baseline over a time-period of 4 hours post-dose (Note that the area only takes values below the individual baseline for the respective visit into account. The area that would result from an increase from baseline is not taken into account for the calculation of the area). Baseline was the last SBP recorded at and within 30 minutes before intake of study drug.
Time Frame: Pre-dose (baseline) and within 4 hours post-dose at visit 6 (week 12)
Population: PD analysis set
Measure: Mean (Standard Deviation); unit: mmHg*h
Arm/Group | Riociguat (Adempas, BAY63-2521) up to 2.5 mg_IDT | Placebo
Number analyzed (Participants) | 10 | 5
mmHg*h | 46.32 (53.57) | 42.44 (28.19)

8. Secondary Outcome: Area Under Effect Curve (AUEC) of Standing SBP Within 4 Hours Post-dose at Visit 6 (Week 12)
Description: The area under effect curve (AUEC) at each visit of standing SBP describes an average within-subject change in SBP from baseline over a time-period of 4 hours post-dose (Note that the area only takes values below the individual baseline for the respective visit into account. The area that would result from an increase from baseline is not taken into account for the calculation of the area). Baseline was the last SBP recorded at and within 30 minutes before intake of study drug.
Time Frame: Pre-dose (baseline) and within 4 hours post-dose at visit 6 (week 12)
Population: PD analysis set
Measure: Mean (Standard Deviation); unit: mmHg*h
Arm/Group | Riociguat (Adempas, BAY63-2521) up to 2.5 mg_IDT | Placebo
Number analyzed (Participants) | 10 | 5
mmHg*h | 38.96 (47.51) | 30.41 (33.35)

9. Secondary Outcome: Area Under Effect Curve (AUEC) of Supine DBP Within 4 Hours Post-dose at Visit 6 (Week 12)
Description: The area under effect curve (AUEC) at each visit of supine DBP describes an average within-subject change in DBP from baseline over a time-period of 4 hours post-dose (Note that the area only takes values below the individual baseline for the respective visit into account. The area that would result from an increase from baseline is not taken into account for the calculation of the area). Baseline was the last DBP recorded at and within 30 minutes before intake of study drug.
Time Frame: Pre-dose (baseline) and within 4 hours post-dose at visit 6 (week 12)
Population: PD analysis set
Measure: Mean (Standard Deviation); unit: mmHg*h
Arm/Group | Riociguat (Adempas, BAY63-2521) up to 2.5 mg_IDT | Placebo
Number analyzed (Participants) | 10 | 5
mmHg*h | 30.79 (35.66) | 32.92 (35.68)

10. Secondary Outcome: Area Under Effect Curve (AUEC) of Standing DBP Within 4 Hours Post-dose at Visit 6 (Week 12)
Description: The area under effect curve (AUEC) at each visit of standing DBP describes an average within-subject change in DBP from baseline over a time-period of 4 hours post-dose (Note that the area only takes values below the individual baseline for the respective visit into account. The area that would result from an increase from baseline is not taken into account for the calculation of the area). Baseline was the last DBP recorded at and within 30 minutes before intake of study drug.
Time Frame: Pre-dose (baseline) and within 4 hours post-dose at visit 6 (week 12)
Population: PD analysis set
Measure: Mean (Standard Deviation); unit: mmHg*h
Arm/Group | Riociguat (Adempas, BAY63-2521) up to 2.5 mg_IDT | Placebo
Number analyzed (Participants) | 10 | 5
mmHg*h | 32.50 (34.04) | 24.20 (22.54)

11. Secondary Outcome: Area Under Effect Curve (AUEC) of Supine HR Within 4 Hours Post-dose at Visit 6 (Week 12)
Description: The area under effect curve (AUEC) at each visit of supine HR describes an average within-subject change in HR from baseline over a time-period of 4 hours post-dose (Note that the area only takes values above the individual baseline for the respective visit into account. The area that would result from a decrease from baseline is not taken into account for the calculation of the area). Baseline was the last HR recorded at and within 30 minutes before intake of study drug.
Time Frame: Pre-dose (baseline) and within 4 hours post-dose at visit 6 (week 12)
Population: PD analysis set
Measure: Mean (Standard Deviation); unit: Beats/min*h
Arm/Group | Riociguat (Adempas, BAY63-2521) up to 2.5 mg_IDT | Placebo
Number analyzed (Participants) | 10 | 5
Beats/min*h | 9.86 (13.08) | 18.85 (14.86)

12. Secondary Outcome: Area Under Effect Curve (AUEC) of Standing HR Within 4 Hours Post-dose at Visit 6 (Week 12)
Description: The area under effect curve (AUEC) at each visit of standing HR describes an average within-subject increase in HR from baseline over a time-period of 4 hours post-dose (Note that the area only takes values above the individual baseline for the respective visit into account. The area that would result from a decrease from baseline is not taken into account for the calculation of the area). Baseline was the last HR recorded at and within 30 minutes before intake of study drug.
Time Frame: Pre-dose (baseline) and within 4 hours post-dose at visit 6 (week 12)
Population: PD analysis set
Measure: Mean (Standard Deviation); unit: Beats/min*h
Arm/Group | Riociguat (Adempas, BAY63-2521) up to 2.5 mg_IDT | Placebo
Number analyzed (Participants) | 10 | 5
Beats/min*h | 13.18 (15.11) | 15.69 (11.81)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected after signing the informed consent until 2 days after end of treatment with the study medication.
Description: Participants completing the main 12-week study phase were allowed to enter a long-term extension phase receiving individual titrated Riociguat at their optimal dose. Long-term extension phase was planned to last until regulatory approval of riociguat but was prematurely terminated by the sponsor.
Arm/Group | Riociguat (Adempas, BAY63-2521) up to 2.5 mg_IDT | Placebo
Serious Adverse Events (participants affected / at risk) | 7/12 | 2/6
Other Adverse Events (participants affected / at risk) | 12/12 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Riociguat (Adempas, BAY63-2521) up to 2.5 mg_IDT (N=12) | Placebo (N=6)
Angina pectoris (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Right ventricular failure (Cardiac disorders) | 1 | 0
Acute right ventricular failure (Cardiac disorders) | 1 | 0
Chronic right ventricular failure (Cardiac disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Erysipelas (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Riociguat (Adempas, BAY63-2521) up to 2.5 mg_IDT (N=12) | Placebo (N=6)
Anaemia (Blood and lymphatic system disorders) | 3 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 0 | 2
Chronic right ventricular failure (Cardiac disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0
Eye swelling (Eye disorders) | 0 | 1
Eyelid oedema (Eye disorders) | 1 | 0
Vision blurred (Eye disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Anal fissure (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 3
Flatulence (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Tongue ulceration (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 2
Epigastric discomfort (Gastrointestinal disorders) | 0 | 1
Regurgitation (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 2 | 0
Chest discomfort (General disorders) | 1 | 0
Chills (General disorders) | 1 | 0
Fatigue (General disorders) | 3 | 0
Oedema (General disorders) | 2 | 1
Oedema peripheral (General disorders) | 7 | 0
Pyrexia (General disorders) | 2 | 1
Inflammation (General disorders) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 2 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 3 | 0
Periodontitis (Infections and infestations) | 1 | 0
Sialoadenitis (Infections and infestations) | 1 | 0
Pharyngotonsillitis (Infections and infestations) | 1 | 0
Peritonitis bacterial (Infections and infestations) | 1 | 0
Oral herpes (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1
Alpha 1 foetoprotein increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 1
Blood bilirubin increased (Investigations) | 1 | 0
Blood cholinesterase decreased (Investigations) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 0
Blood potassium decreased (Investigations) | 0 | 2
Blood pressure systolic decreased (Investigations) | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1
Glomerular filtration rate decreased (Investigations) | 1 | 0
Lymphocyte count decreased (Investigations) | 1 | 0
Neutrophil count increased (Investigations) | 1 | 0
Weight decreased (Investigations) | 0 | 1
Glutamate dehydrogenase increased (Investigations) | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Iron deficiency (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 4 | 2
Headache (Nervous system disorders) | 3 | 3
Sciatica (Nervous system disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Renal failure chronic (Renal and urinary disorders) | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Cataract operation (Surgical and medical procedures) | 1 | 0
Capillary fragility (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 6 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The embargo can be up to 6 months (equal to the 180 days), moreover if it is necessary the embargo period can be prolonged to expiry of priority year.